CLINICAL TRIAL: NCT01971164
Title: Randomized, Single-blind, Placebo-controlled, Multiple Ascending Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics & Pharmacodynamics of JTZ-951 Administered Once Daily for 15 Days in Anemic Subjects With End-stage Renal Disease
Brief Title: Safety, Tolerability, PK & PD Study of JTZ-951 in Anemic Subjects With End-stage Renal Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AZ951-U-12-004
Record Dates: First submitted 2013-10-15; First posted 2013-10-29 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: anemia; chronic kidney disease; hemodialysis
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — enarodustat

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose 1 JTZ-951 or Placebo (Experimental): Tablets, 1 dose per day for 15 days
  Interventions: Drug: JTZ-951; Drug: Placebo
- Dose 2 JTZ-951 or Placebo (Experimental): Tablets, 1 dose per day for 15 days
  Interventions: Drug: JTZ-951; Drug: Placebo
- Dose 3 JTZ-951 or Placebo (Experimental): Tablets, 1 dose per day for 15 days
  Interventions: Drug: JTZ-951; Drug: Placebo
- Dose 4 JTZ-951 or Placebo (Experimental): Tablets, 1 dose per day for 15 days
  Interventions: Drug: JTZ-951; Drug: Placebo

INTERVENTIONS:
Drug: JTZ-951 — Subjects will receive JTZ-951 or Placebo
Drug: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of sequential ascending doses of JTZ-951 administered for 15 days in anemic subjects with end-stage renal disease (ESRD) receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have ESRD and have been receiving maintenance hemodialysis for at least 12 weeks prior to the Screening Visit
* Body weight (post-dialysis weight) greater than 45.0 kg and a body mass index between 20.0 and 40.0 kg/m2 (inclusive) at the Screening Visit
* Hemoglobin value as defined in the protocol
* Meet the erythropoiesis-stimulating agent (ESA) therapy criteria at the Screening Visit as defined in the protocol

Exclusion Criteria:

* Transferrin saturation and ferritin levels at the Screening Visit as defined in the protocol
* Anemia due to known causes other than chronic kidney disease
* Known history of hyporesponsiveness to ESAs
* Acute coronary syndrome (e.g., myocardial infarction) within 1 year prior to Screening visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | 15 days
Vital signs and 12 lead ECGs | 15 days
Cmax (maximum concentration) | 15 days
tmax (time to reach maximum concentration) | 15 days
t1/2 (elimination half-life) | 15 days
AUC (area under the concentration-time curve) | 15 days
AR (accumulation ratio) | 15 days
RBC (red blood cell) count | 15 days
Hgb (hemoglobin) | 15 days
TSAT (transferrin saturation) | 15 days
serum ferritin | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Hideyuki Yamamoto, Study Chair — Akros Pharma Inc.
Locations (5):
- United States (5):
  - Lakewood, Colorado
  - Miami, Florida
  - Orlando, Florida
  - Minneapolis, Minnesota
  - Saint Paul, Minnesota

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278